CLINICAL TRIAL: NCT00821015
Title: Effect of Balloon Cryoablation on Left Atrial Function (CRYO-LA)
Brief Title: Effect of Balloon Cryoablation on Left Atrial Function
Acronym: CRYO-LA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, DIRECTOR CARDIAC ARRHYTHMIA SERVICE, PROFESSOR OF MEDICINE, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 09-0628
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
Keywords: cryoablation; recurring arrhythmia; stroke; RF ablation; LA ablation; nodal ablation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- Experimental (Experimental): All study subjects will undergo cryoablation. This is a non-randomized trial.
  Interventions: Device: Pulmonary vein isolation with cryoballoon catheter

INTERVENTIONS:
Device: Pulmonary vein isolation with cryoballoon catheter — For each patient, the balloon catheter will be advanced to the ostium of each pulmonary vein. Once location has been optimized, the balloon will be inflated, and cryoenergy delivery will be initiated. Because the entire surface of the balloon acts as an ablative surface, circumferential ablation of each pulmonary vein will be achieved concurrently. This will be completed for each pulmonary vein for each patient.

SUMMARY:
Atrial fibrillation is a common and disabling irregular heart rhythm, that affects 1 to 1.5 million Americans. Recent clinical experience with the Medtronic Arctic Front™ Cardiac CryoAblation Catheter System suggests that it can be used to isolate the pulmonary veins (PVs) safely and effectively in patients with AF, thereby reducing or eliminating the recurrence of AF.3-4 However, the very large ablative surface of this balloon ablation catheter raises the possibility that this technique may damage extensive areas of the atrial myocardium.

The LA is an elastic chamber, designed to expand and contract with ease to accommodate the influx and outflow of blood, while maintaining relatively low pressure. When exposed to stress or injury, whether acute or chronic, the LA may lose much of its elasticity, resulting in overall dilation accompanied by fibrosis in some cases. Overall, this may potentially result in diminution of LA mechanical function (both systolic contractile function, and diastolic relaxation function). In addition, LA function is linked to both Left Ventricular (LV) systolic and diastolic function, manifesting in an overall impact on cardiac remodeling, including the area of the pulmonary vein ostia, and a significant decrease in LV ejection fraction (LVEF). On the other hand, the positive effects of maintaining sinus rhythm with successful catheter ablation of AF may result in improvement of LA mechanical function.5-9

Based on the potentially deleterious effects of damage caused by cryoablation, to the atrial myocardium during balloon ablation, this prospective, non-randomized, single-center study has been designed to assess the atrial effects of balloon cryo-ablation.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, single-center, controlled study of patients with AF referred for ablation after failing one or more Class I-IV antiarrhythmic drugs used in the treatment of AF.

• All study subjects will undergo cryoablation.

Subjects will be followed for 12 months to assess the chronic impact of ablation with the Medtronic CryoCath Arctic Front™ Cardiac CryoAblation Catheter System on LA and LV mechanical function. In addition, patients will undergo scheduled and symptom-driven assessments to detect recurrent AF and adverse events (AEs).

We will evaluate the effect of ablation with the Medtronic Arctic Front™ Cardiac CryoAblation Catheter System on the atrial myocardium, with respect to LA (and LV) mechanical function, by assessing images acquired using TTE and CT in adult patients with atrial fibrillation who have failed at least one anti-arrhythmic drug. The efficacy of the Arctic Front™ Cardiac CryoAblation Catheter System will be assessed by ambulatory continuous ECG monitoring

ELIGIBILITY:
Inclusion Criteria:

* Documented paroxysmal atrial fibrillation
* ≥ 18 and ≤ 85 years of age
* Failure of one or more AF Drugs (AFDs).
* Referral for a pulmonary vein isolation catheter ablation procedure to treat atrial fibrillation
* Ability to understand the requirements of the study
* Willingness to adhere to study restrictions and comply with all post- procedural follow-up requirements

Exclusion Criteria:

* Any reversible cause of AF (post-surgery, thyroid disorder, etc.)
* More than 4 cardioversions in the prior year.
* Patients with recent myocardial infarction (less than 2 months) or unstable angina.
* Patients with congestive heart failure (NYHA class III or IV).
* Patients who have experienced any cerebral ischemic event, including any TIA in the preceding 1 month.
* Women who are known to be pregnant or have had a positive β-HCG test 7 days prior to procedure.
* Patients with any other significant uncontrolled or unstable medical condition (including uncontrolled clinically significant coagulation disorders).
* Patients whose life expectancy is less than one year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Y Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for the Management of Patients with Atrial Fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Aug 15;114(7):e257-354. doi: 10.1161/CIRCULATIONAHA.106.177292. No abstract available. PMID 16908781
- [Background] European Heart Rhythm Association (EHRA); European Cardiac Arrhythmia Scoiety (ECAS); American College of Cardiology (ACC); American Heart Association (AHA); Society of Thoracic Surgeons (STS); Calkins H, Brugada J, Packer DL, Cappato R, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, Haines DE, Haissaguerre M, Iesaka Y, Jackman W, Jais P, Kottkamp H, Kuck KH, Lindsay BD, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Natale A, Pappone C, Prystowsky E, Raviele A, Ruskin JN, Shemin RJ. HRS/EHRA/ECAS expert Consensus Statement on catheter and surgical ablation of atrial fibrillation: recommendations for personnel, policy, procedures and follow-up. A report of the Heart Rhythm Society (HRS) Task Force on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2007 Jun;4(6):816-61. doi: 10.1016/j.hrthm.2007.04.005. Epub 2007 Apr 30. No abstract available. PMID 17556213
- [Background] Reddy VY, Neuzil P, d'Avila A, Laragy M, Malchano ZJ, Kralovec S, Kim SJ, Ruskin JN. Balloon catheter ablation to treat paroxysmal atrial fibrillation: what is the level of pulmonary venous isolation? Heart Rhythm. 2008 Mar;5(3):353-60. doi: 10.1016/j.hrthm.2007.11.006. Epub 2007 Nov 7. PMID 18313591
- [Background] Van Belle Y, Janse P, Rivero-Ayerza MJ, Thornton AS, Jessurun ER, Theuns D, Jordaens L. Pulmonary vein isolation using an occluding cryoballoon for circumferential ablation: feasibility, complications, and short-term outcome. Eur Heart J. 2007 Sep;28(18):2231-7. doi: 10.1093/eurheartj/ehm227. Epub 2007 Jun 14. PMID 17569680
- [Background] Tsao HM, Wu MH, Huang BH, Lee SH, Lee KT, Tai CT, Lin YK, Hsieh MH, Kuo JY, Lei MH, Chen SA. Morphologic remodeling of pulmonary veins and left atrium after catheter ablation of atrial fibrillation: insight from long-term follow-up of three-dimensional magnetic resonance imaging. J Cardiovasc Electrophysiol. 2005 Jan;16(1):7-12. doi: 10.1046/j.1540-8167.2005.04407.x. PMID 15673379
- [Background] Lemola K, Desjardins B, Sneider M, Case I, Chugh A, Good E, Han J, Tamirisa K, Tsemo A, Reich S, Tschopp D, Igic P, Elmouchi D, Bogun F, Pelosi F Jr, Kazerooni E, Morady F, Oral H. Effect of left atrial circumferential ablation for atrial fibrillation on left atrial transport function. Heart Rhythm. 2005 Sep;2(9):923-8. doi: 10.1016/j.hrthm.2005.06.026. PMID 16171744
- [Background] Verma A, Kilicaslan F, Adams JR, Hao S, Beheiry S, Minor S, Ozduran V, Claude Elayi S, Martin DO, Schweikert RA, Saliba W, Thomas JD, Garcia M, Klein A, Natale A. Extensive ablation during pulmonary vein antrum isolation has no adverse impact on left atrial function: an echocardiography and cine computed tomography analysis. J Cardiovasc Electrophysiol. 2006 Jul;17(7):741-6. doi: 10.1111/j.1540-8167.2006.00488.x. PMID 16836670
- [Background] Reant P, Lafitte S, Jais P, Serri K, Weerasooriya R, Hocini M, Pillois X, Clementy J, Haissaguerre M, Roudaut R. Reverse remodeling of the left cardiac chambers after catheter ablation after 1 year in a series of patients with isolated atrial fibrillation. Circulation. 2005 Nov 8;112(19):2896-903. doi: 10.1161/CIRCULATIONAHA.104.523928. Epub 2005 Oct 31. PMID 16260634
- [Background] Yamanaka K, Fujita M, Doi K, Tsuneyoshi H, Yamazato A, Ueno K, Zen E, Komeda M. Multislice computed tomography accurately quantifies left atrial size and function after the MAZE procedure. Circulation. 2006 Jul 4;114(1 Suppl):I5-9. doi: 10.1161/CIRCULATIONAHA.105.000968. PMID 16820627

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects presenting with AF for ablation recruited from the clinical practice of the Investigators.
Groups:
- Cryoballoon Catheter: All study subjects will undergo cryoablation. This is a non-randomized trial.
  Pulmonary vein isolation with cryoballoon catheter: For each patient, the balloon catheter will be advanced to the ostium of each pulmonary vein. Once location has been optimized, the balloon will be inflated, and cryoenergy delivery will be initiated. Because the entire surface of the balloon acts as an ablative surface, circumferential ablation of each pulmonary vein will be achieved concurrently. This will be completed for each pulmonary vein for each patient.
Period: Overall Study
Arm/Group | Cryoballoon Catheter
Started | 27
Completed | 15
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 17
Height [Mean (Standard Deviation); unit: inches] | 68.2 (4.22)
Weight [Mean (Standard Deviation); unit: pounds] | 183.5 (40.8)
Participants with Risk Factors [Count of Participants; unit: Participants]
  Diabetes | 1
  Hypertension | 13
  Smoking | 3
  Alcohol Abuse | 0
  Coronary Artery Disease | 4
  Myocardial Infarction | 2
Atrial Flutter [Count of Participants; unit: Participants] — Arrhythmia History - Atrial flutter
  Participants | 5
Number of Prior Cardioversions [Mean (Standard Deviation); unit: cardioversions] | .66 (.09)
Number of Hospital Admissions for AF [Mean (Standard Deviation); unit: hospital admissions] | .22 (.08)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Procedural Success (APS)
Description: Acute Procedural Success (APS) is the demonstration of electrical isolation of all 4 PVs or their anomalous equivalents at the conclusion of the first protocol-defined cryoablation procedure.
Time Frame: Immediately following procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 27
Participants | 27

2. Primary Outcome: Number of Participants With AF Recurrence
Description: Number of Participants with AF Recurrence at 6 months and at 12 months after Cryoballoon Ablation for Atrial Fibrillation.
  (Chronic Treatment Success is defined as a subject who does not have episodes of AF, lasting at least 30 seconds in duration, 3 months following the initial ablation procedure.)
Time Frame: 6 months and 12 months
Population: Only subjects who returned for their visit was included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 26
Participants
  6 months | 3
  12 months: number analyzed (Participants) | 19
  12 months | 1

3. Primary Outcome: Left Atrial Measurements
Description: Transthoracic Echo Assessment of Left Atrial Function at Baseline and 6-Months Post- Cryoballoon Ablation for AF
  Parameters of atrial function:
  1. Volumes at P-wave onset and end-systole
  2. LA active emptying volume
  3. LA active emptying fraction
  4. Late diastolic peak velocity
  5. LA filling fraction
  6. Pulmonary venous inflow pattern
Time Frame: Baseline and 6 months
Population: Echocardiogram data was incomplete for 9 patients.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 18
cm
  Parasternal baseline | 3.79 (0.55)
  Parasternal 6 months | 3.77 (0.54)
  Longitudinal baseline | 5.70 (0.72)
  Longitudinal 6 months | 5.33 (0.9)
  Transverse baseline | 4.21 (0.61)
  Transverse 6 months | 3.82 (0.95)

4. Primary Outcome: LVEF
Description: Ventricular Function measured by Left Ventricular Ejection Function (LVEF). A normal left ventricular ejection fraction (LVEF) ranges from 55% to 70%. An LVEF of 65%, for example means that 65% of total amount of blood in the left ventricle is pumped out with each heartbeat.
Time Frame: Baseline and 6 months
Population: Echocardiogram data was incomplete for 9 patients.
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 18
percentage of blood
  Baseline | 59 (0.05)
  6 months | 62 (0.09)

5. Primary Outcome: Left Atrial Volume
Description: Transthoracic Echo Assessment of Left Atrial Function at Baseline and 6-Months Post- Cryoballoon Ablation for AF
Time Frame: Baseline and 6 months
Population: Echocardiogram data was incomplete for 9 patients.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 18
ml
  End-Systolic Volume baseline | 60.62 (11.9)
  End-Systolic Volume 6 months | 54.71 (36.08)
  Pre-P Volume baseline: number analyzed (Participants) | 15
  Pre-P Volume baseline | 36.87 (13.0)
  Pre-P Volume 6 months: number analyzed (Participants) | 15
  Pre-P Volume 6 months | 33.63 (16.37)
  End-Diastolic Volume baseline | 25.69 (24.12)
  End-Diastolic Volume 6 months | 24.08 (54.69)

6. Primary Outcome: Deflections of the Mitral Annulus Measurement
Description: Transthoracic Echo Assessment of Left Atrial Function at Baseline and 6-Months Post- Cryoballoon Ablation for AF Deflections of the mitral annulus as measured by peak early ventricular diastolic velocity (E'), and during atrial contraction (A')
Time Frame: Baseline and 6 months
Population: Echocardiographic data was incomplete for 9 participants
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 18
cm/s
  E at baseline | 64.00 (16.75)
  E at 6 months | 64.82 (13.68)
  A at baseline: number analyzed (Participants) | 15
  A at baseline | 58.95 (17.34)
  A at 6 months: number analyzed (Participants) | 15
  A at 6 months | 54.18 (14.04)

7. Secondary Outcome: Chronic Treatment Success for the Follow-up Visit Within Treatment Windows.
Description: Chronic Treatment Success for the follow-up visit within treatment windows. 1. Whether on or off Atrial Fibrillation Drugs (AFDs) during the Non-blanked Follow-up Period 2. When off Atrial Fibrillation Drugs
Time Frame: 3 months
Population: Data about atrial fibrillation drugs during the 3 month period were unfortunately not collected for any participant in the study for this outcome measure.
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 0

8. Secondary Outcome: Atrial Flutter
Description: 1. Flutter Acute Procedural Success 2. Freedom from Flutter Chronic Treatment Failure
Time Frame: 3 months
Population: Data about atrial flutter procedural success were not collected for any participant in the study for this outcome measure.
Arm/Group | Cryoballoon Catheter
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cryoballoon Catheter
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27
Other Adverse Events (participants affected / at risk) | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoballoon Catheter (N=27)
Central Retinal Artery Occlusion (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes